CLINICAL TRIAL: NCT04936594
Title: Transcranial Magnetic Stimulation (TMS) for Smoking Cessation in People Living With HIV/AIDS (PLWHA)
Brief Title: TMS for Smoking Cessation in PLWHA Cessation in People Living With HIV/AIDS (PLWHA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gopalkumar Rakesh (Other)
Responsible Party: Sponsor-Investigator, Gopalkumar Rakesh, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 64473
Record Dates: First submitted 2021-06-02; First posted 2021-06-23 (Actual); Results first posted 2023-07-13 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-06

CONDITIONS: Smoking Cessation; HIV; Craving
Keywords: Transcranial magnetic stimulation (TMS); Attentional bias; Conditioning
MeSH Terms: conditions — Smoking Cessation | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Single blind within participant design
Masking Description: All participants received iTBS (intermittent theta burst stimulation) first and sham subsequently but were blinded regarding treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- People Living with HIV/AIDS Who Smoke (Experimental): Participants will be people living with HIV/AIDS who smoke. They will receive two interventions: iTBS and a sham comparator (TMS).
  Interventions: Device: iTBS; Device: TMS

INTERVENTIONS:
Device: iTBS — 1800 pulses of iTBS
  Other Names: Intermittent theta burst stimulation
Device: TMS — MagVenture MagPro x100 device. This will be used as the comparator.
  Other Names: Transcranial magnetic stimulation

SUMMARY:
The pilot study proposal aims to modulate craving and attentional bias towards smoking cues in 40 people living with HIV/AIDS (PLWHA) using transcranial magnetic stimulation (TMS), with functional MRI (fMRI) brain correlates. TMS is a form of noninvasive brain stimulation and modulates neural activity using tiny doses of focused electricity. For the study, participants would perform two cognitive tasks and neuroimaging before and after the TMS and investigators would compare changes in these paradigms with TMS. The investigators will also get a point of contact urine drug screen before study initiation. The investigators will aim to recruit 20 subjects in each arm of our trial (total of 40) from the BlueGrass HIV Clinic.

DETAILED DESCRIPTION:
People living with HIV/AIDS (PLWHA) smoke at nearly three times the rate of the general population. These extraordinary smoking rates are associated with greater AIDS-related cancer, non-AIDS related morbidity including non-AIDS-defining cancer, cardiovascular disease, pulmonary disease, and mortality. Smoking significantly impacts the progression and outcome of HIV disease and has been identified as the leading contributor to premature mortality in PLWHA. Suboptimal results with current smoking cessation strategies makes identifying new adjunct strategies an area of need. The pilot study proposal aims to modulate craving and attentional bias towards smoking cues in people living with HIV/AIDS (PLWHA) using transcranial magnetic stimulation (TMS), with functional MRI (fMRI) brain correlates. TMS is a form of noninvasive brain stimulation and modulates neural activity using tiny doses of focused electricity. The TMS paradigm we would be performing is called theta burst stimulation (TBS), which is potent, short, and efficient. It has shown to cause neuroplasticity even with a single session and was approved by the FDA for treatment of major depressive disorder in 2019.

Targeting the left dorsolateral prefrontal cortex (DLPFC) by using MNI coordinates (-44,40,29) via Brainsight Neuronavigation will modulate craving and attentional bias that is closely associated with craving. For this pilot study, 40 participants will perform the attentional bias task, craving scale and neuroimaging before and after the TBS/ sham TMS session, to compare changes in these paradigms between these interventions. Attentional bias would be measured with eye tracking, craving will be assessed with tobacco craving questionnaire (TCQ-SF). The investigators will aim to recruit 10 subjects from the BlueGrass HIV Clinic, who have an established pipeline for enrolling PLWHA patients in clinical trials. Although there is limited data on TMS in smoking, there have been no TMS studies done in PLWHA

ELIGIBILITY:
Inclusion Criteria:

* Patients enrolled in the Bluegrass Clinic
* Confirmed chart diagnosis of a HIV and receiving HIV treatment at the participating HIV clinic
* Age 18-60 years
* Preferably right hand dominant
* Currently self-report smoking 10 of more cigarettes per day or a score of > 5 on the Fagerstrom Test for Nicotine
* Willing and able to abstain from all drug use
* Exhaled breath on day of study Carbon Monoxide < 10 ppm
* Stabilized on maintenance buprenorphine if having comorbid opioid use disorder
* Able to read and speak English
* Able to provide informed consent to participate.

Exclusion Criteria:

* Pregnant, nursing, or becoming pregnant during the study
* History of traumatic brain injury or seizures which are contraindications for transcranial magnetic stimulation (TMS)
* Increased risk of seizure for any reason, including prior diagnosis of epilepsy, seizure disorder, increased intracranial pressure, or history of significant head trauma with loss of consciousness for ≥ 5 minutes which are all contraindications for TMS
* Presence of intracranial implants (e.g. aneurysms clips, shunts, stimulators, cochlear implants, or electrodes), cardiac pacemakers, or vagus nerve stimulation device which are all contraindications for magnetic resonance imaging
* Neurological disorder including, but not limited to: space occupying brain lesion; any history of seizures, history of cerebrovascular accident; fainting, cerebral aneurysm, major neurocognitive disorder, Huntington chorea; multiple sclerosis which are all contraindications for TMS.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2021-05-24 (Actual); Primary Completion 2021-11-24 (Actual); Study Completion 2021-11-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gopalkumar Rakesh, MD, Principal Investigator — Assistant Professor, University of Kentucky
Locations (1):
- 245 Fountain Court, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 9 participants were enrolled; however, 1 participant dropped out before the experimental sessions began.
Groups:
- People Living With HIV/AIDS Who Smoke: Participants will be people living with HIV/AIDS who smoke. They will receive two interventions: iTBS (Intermittent Theta Burst Stimulation) and a sham comparator (TMS).
Period: Overall Study
Arm/Group | People Living With HIV/AIDS Who Smoke
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | People Living With HIV/AIDS Who Smoke
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.88 (3.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Change in Attentional Bias iTBS (Intermittent Theta Burst Stimulation) Smoking
Description: Cues Encompassing People Smoking Cigarettes. Measured after iTBS using visual probe task administered (adapted for smoking images) on a computer and eye tracker. Images of smoking and a matched neutral cue were presented on a laptop screen, 3 cm apart. Upon offset of the image pairs, a visual probe (X) appeared on either the left side or right side of the screen, in the same location as one of the previously presented images. Attentional bias is quantified using fixation time on cigarette and neutral cues, via an eye tracker in milliseconds
Time Frame: baseline and immediately after intervention, approximately 4 hours
Measure: Mean (Standard Error); unit: milliseconds
Groups:
- People Living With HIV/AIDS (PLWHA) Who Smoke: Participants will be people living with HIV/AIDS who smoke. They will receive two interventions: iTBS and a sham comparator (TMS).
Arm/Group | People Living With HIV/AIDS (PLWHA) Who Smoke
Number analyzed (Participants) | 8
milliseconds
  Baseline | 1007.05 (148.70)
  After Intervention | 566.89 (121.70)

2. Primary Outcome: Change in Attentional Bias Sham Smoking
Description: Cues Encompassing People Smoking Cigarettes. Measured after sham using visual probe task (adapted for smoking images) administered on a computer and eye tracker. Images of smoking and a matched neutral cue were presented on a laptop screen, 3 cm apart. Upon offset of the image pairs, a visual probe (X) appeared on either the left side or right side of the screen, in the same location as one of the previously presented images. Attentional bias is quantified using fixation time on cigarette and neutral cues, via an eye tracker in milliseconds
Time Frame: baseline and immediately after intervention, approximately 4 hours
Population: 3 participants who got itbs did not show up for the sham visit
Measure: Mean (Standard Error); unit: milliseconds
Arm/Group | People Living With HIV/AIDS Who Smoke
Number analyzed (Participants) | 5
milliseconds
  Baseline | 884.60 (112.77)
  After Intervention | 658.67 (148.63)

3. Primary Outcome: Change in Attentional Bias iTBS Paraphernalia
Description: Cues Encompassing Cigarette Paraphernalia. Measured after iTBS using visual probe task (adapted for smoking images) administered on a computer and eye tracker. Images of cigarette paraphernalia and a matched neutral cue were presented on a laptop screen, 3 cm apart. Upon offset of the image pairs, a visual probe (X) appeared on either the left side or right side of the screen, in the same location as one of the previously presented images. Attentional bias is quantified using fixation time on cigarette and neutral cues, via an eye tracker in milliseconds
Time Frame: baseline and immediately after intervention, approximately 4 hours
Measure: Mean (Standard Error); unit: milliseconds
Arm/Group | People Living With HIV/AIDS Who Smoke
Number analyzed (Participants) | 8
milliseconds
  Baseline | 670.43 (139.26)
  After Intervention | 443.10 (136.37)

4. Primary Outcome: Change in Attentional Bias Sham Paraphernalia
Description: Cues Encompassing Cigarette Paraphernalia. Measured after sham using visual probe task (adapted for smoking images) administered on a computer and eye tracker. Images of cigarette paraphernalia and a matched neutral cue were presented on a laptop screen, 3 cm apart. Upon offset of the image pairs, a visual probe (X) appeared on either the left side or right side of the screen, in the same location as one of the previously presented images. Attentional bias is quantified using fixation time on cigarette and neutral cues, via an eye tracker in milliseconds
Time Frame: baseline and immediately after intervention, approximately 4 hours
Population: 3 participants who got itbs did not show up for the sham visit
Measure: Mean (Standard Error); unit: milliseconds
Arm/Group | People Living With HIV/AIDS Who Smoke
Number analyzed (Participants) | 5
milliseconds
  Baseline | 528.38 (139.39)
  After Intervention | 307.56 (135.26)

5. Secondary Outcome: Change in Tobacco Craving Questionnaire Short Form (TCQ-SF) iTBS
Description: Craving measured using TCQ-SF. The Tobacco Craving Questionnaire-short form (TCQ-SF) consists of 12 items rated on a visual analogue scale from 0 to 84 with a higher score equating to increased craving.
Time Frame: baseline and immediately after intervention, approximately 4 hours
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | People Living With HIV/AIDS Who Smoke
Number analyzed (Participants) | 8
score on a scale
  Baseline | 55.88 (3.95)
  After Intervention | 43.13 (4.68)

6. Secondary Outcome: Change in Tobacco Craving Questionnaire Short Form (TCQ-SF) Sham
Description: as for outcome 5
Time Frame: baseline and immediately after intervention, approximately 4 hours
Population: All participants completed the iTBS session but 3 participants did not show up for the sham visit
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | People Living With HIV/AIDS Who Smoke
Number analyzed (Participants) | 5
score on a scale
  Baseline | 53.2 (4.77)
  After Intervention | 48.40 (6.84)

7. Other Pre Specified Outcome: Resting State Functional Connectiivity
Description: Measured in MRI scanner
Time Frame: Baseline
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Resting State Functional Connectiivity
Description: Measured in MRI scanner
Time Frame: Four hours from baseline
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 4 weeks after intervention
Arm/Group | People Living With HIV/AIDS (PLWHA) Who Smoke
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-02-07): https://cdn.clinicaltrials.gov/large-docs/94/NCT04936594/Prot_SAP_ICF_000.pdf